CLINICAL TRIAL: NCT04411849
Title: A Multilevel HPV Self-Testing Intervention to Increase Cervical Cancer Screening Among Women in Appalachia
Brief Title: Multilevel HPV Self-Testing Intervention for the Increase of Cervical Cancer Screening Among Women in Appalachia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Paul Reiter, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: OSU-20055; NCI-2020-01228 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P01CA229143 (NIH)
Record Dates: First submitted 2020-05-28; First posted 2020-06-02 (Actual); Results first posted 2024-12-04 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Cervical Carcinoma; Human Papillomavirus Infection
MeSH Terms: conditions — Uterine Cervical Neoplasms; Papillomavirus Infections | interventions — Practice Guidelines as Topic; Standard of Care; Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (intervention) (Experimental): Participants receive the HPV self-testing intervention consisting of mailed HPV self-test devices. Participants also receive an information about cervical cancer. Participants who do not return their self-test within a few weeks receive telephone-based patient navigation.
  Interventions: Procedure: HPV Self-Collection; Other: Informational Intervention; Behavioral: Patient Navigation Program
- Group II (usual care continued) (Active Comparator): Participants receive usual care consisting of a reminder letter to get a clinic-based cervical cancer screening test and information about cervical cancer.
  Interventions: Other: Best Practice; Other: Informational Intervention

INTERVENTIONS:
Other: Best Practice — Receive usual care
  Other Names: standard of care; standard therapy
  Arms: Group II (usual care continued)
Procedure: HPV Self-Collection — Receive HPV self-testing intervention
  Other Names: At-home HPV Self Collection; HPV Self Collection; Human Papillomavirus Self-Collection
  Arms: Group I (intervention)
Other: Informational Intervention — Receive information about cervical cancer
Behavioral: Patient Navigation Program — Receive telephone-based patient navigation
  Other Names: Patient Navigator Program
  Arms: Group I (intervention)

SUMMARY:
This trial studies how well a multilevel human papillomavirus (HPV) self-testing intervention works in increasing cervical cancer screening among women in Appalachia. Most cases of cervical cancer occur among unscreened and underscreened women. A multilevel HPV self-testing intervention may help to improve cervical cancer screening rates.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

Determine the effectiveness of the intervention in increasing cervical cancer screening.

OUTLINE: Participants are randomized to 1 of 2 groups.

GROUP I: Participants receive the HPV self-testing intervention consisting of mailed HPV self-test devices. Participants also receive an information about cervical cancer. Participants who do not return their self-test within a few weeks receive telephone-based patient navigation.

GROUP II: Participants receive usual care consisting of a reminder letter to get a clinic-based cervical cancer screening test and information about cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* Not within recommended cervical cancer screening guidelines for women in this age range (i.e., no Papanicolaou [Pap] test in last 3 years or no Pap test plus clinic-based HPV test in last 5 years)
* Resident of an Appalachian county
* Not currently pregnant
* Intact cervix
* No history of invasive cervical cancer
* Seen in a participating clinic/health system in last 2 years (i.e., active patient)
* Have a working telephone

Ages: 30 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 802 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2024-06-11 (Actual); Study Completion 2024-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Reiter, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (4):
- United States (4):
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Virginia, Charlottesville, Virginia
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Group I (Intervention): Participants receive the HPV self-testing intervention consisting of mailed HPV self-test devices. Participants also receive an information about cervical cancer. Participants who do not return their self-test within a few weeks receive patient navigation.
  HPV Self-Collection: Receive HPV self-testing intervention
  Informational Intervention: Receive information about cervical cancer
  Patient Navigation Program: Receive patient navigation
Period: Overall Study
Arm/Group | Group I (Intervention) | Group II (Usual Care Continued)
Started | 464 | 338
Completed | 464 | 338
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I (Intervention) | Group II (Usual Care Continued) | Total
Number analyzed (Participants) | 464 | 338 | 802
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 464 | 338 | 802
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 464 | 338 | 802
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 464 | 338 | 802

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness of Human Papillomavirus (HPV) Intervention
Description: The patient-level effectiveness will be whether or not women get "screened" during the project. Will examine the proportion of women screened, and use an intent-to-treat approach. To compare treatment groups (Group 1 versus Group 2), will use generalized linear mixed models (GLMMs) to account for the correlation between women from the same health system.
Time Frame: Up to 1 years
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Intervention) | Group II (Usual Care Continued)
Number analyzed (Participants) | 464 | 338
Participants | 69 | 17

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Group I (Intervention) | Group II (Usual Care Continued)
All-Cause Mortality (participants affected / at risk) | 0/464 | 0/338
Serious Adverse Events (participants affected / at risk) | 0/464 | 0/338
Other Adverse Events (participants affected / at risk) | 0/464 | 0/338

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-30): https://cdn.clinicaltrials.gov/large-docs/49/NCT04411849/Prot_SAP_000.pdf